CLINICAL TRIAL: NCT01171638
Title: The Use of Near Infrared Spectroscopy in the Diagnosis of Acute Compartment Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: J&M Shuler (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Nonin Medical (Unknown)
Responsible Party: Brett Freedman, MAJ MC (MD), Landstuhl Regional Medical Center
Other Study IDs: DR080018-02
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Acute Compartment Syndrome
Keywords: near infrared spectroscopy; compartment syndrome; fasciotomy; INVOS
MeSH Terms: conditions — Compartment Syndromes | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Critical Controls: Critically injured patients with NO "severe traumatic lower extremity" injuries to provide normative data for the "critically injured" physiological status upon arrival at study site
  Interventions: Device: Near infrared spectroscopy (NIRS)
- Investigational cohort: Soldiers with "severe traumatic lower extremity" injuries in "stable" or "critical" physiological status presenting to a participating study site within 12 hours of their injury, to provide data on the acute post-injury phase. This cohort will be made up of:
  * Patients meeting inclusion criteria for investigational cohort, who have UNILATERAL "severe lower extremity injuries"
  * Patients meeting inclusion criteria for investigational cohort, who have BILATERAL "severe lower extremity injuries."
  * Patients meeting inclusion criteria for investigational cohort, who have been clinically diagnosed by the treating provider using that treating providers standards for diagnosing ACS and the patient in addition to be diagnosed with ACS undergoes four-compartment leg fasciotomy.
  Interventions: Device: Near infrared spectroscopy (NIRS)

INTERVENTIONS:
Device: Near infrared spectroscopy (NIRS) — Non-invasive monitoring device applied on the surface of the skin that emits harmless red light to measure tissue perfusion.
  Other Names: Equanox Regional Oximeter, Nonin Medical, Plymouth, MN

SUMMARY:
This is a prospective observational study to determine the reliability and accuracy of Near Infrared Spectroscopy (NIRS) to detect oxygen flow in the extremities of injured and non-injured soldiers over time. This technology may be useful in the detection of acute compartment syndrome. We hypothesize that:

* NIRS values will be well-correlated with intracompartmental pressure measurements
* NIRS values will be significantly different between non-injured and injured extremities, and injured extremities treated with fasciotomy for acute compartment syndrome.
* NIRS values of the upper extremity and feet will correlate to values from normal legs in critical control patients and patients with unilateral sever lower extremity injuries.

DETAILED DESCRIPTION:
The purpose of this prospective observational cohort study is to define the reliability and accuracy of Near Infrared Spectroscopy (NIRS) in the detection of intra-compartmental tissue perfusion in injured and noninjured extremities over time. Additionally, it will establish diagnostic perfusion value thresholds to be used in a subsequent interventional study confirming the efficacy of NIRS-based ACS monitoring. Through prospective measurements of NIRS values, vital signs, intracompartmental pressures and clinical examinations, guidelines and parameters will be established for the use of NIRS in diagnosing acute compartment syndrome (ACS), monitoring patients at risk for ACS and evaluating the adequacy of fasciotomy in patients treated for ACS.

Null hypotheses:

* NIRS values do not correlate with intracompartmental pressures, when they are obtained in the course of routine care of patients in the combat theater.
* There is no difference in the NIRS values between non-injured, injured extremities and injured extremities treated with fasciotomy for ACS
* NIRS values from the upper extremity and feet do not correlate to NIRS values from the normal legs in critical control patients and patients with unilateral severe lower extremity injury.

Specific Aims:

1. Conduct observational, human-use, study to compile a normative reference database for NIRS-measured tissue perfusion in the uninjured upper extremity and the injured and non-injured legs of up to 120 injured subjects, from varying ethnicities (skin pigmentations) in varying degrees of hemodynamic status (stable, critically injured) to test the 3 hypotheses listed above. The study groups consist of one control group (critically ill without leg injuries) and one investigational group (critically injured with leg injuries):

   * COHORT 1: 25 critically injured patients with NO severe traumatic lower extremity traumatic injuries to provide normative data for the "critically injured" physiological status ("Critical" CONTROLS)
   * COHORT 2: 95 total (35 Cohort 2A; 35 Cohort 2B; 25 Cohort 2C) patients with "severe" traumatic lower extremity injuries presenting to a "participating" level 1 trauma center within 12 hours of their injury, to provide data on the acute post-injury phase. (INVESTIGATIONAL COHORT)
   * COHORT 2A: Patients meeting COHORT 2 inclusion criteria, who have UNILATERAL "severe lower extremity injuries".
   * COHORT 2B: Patients meeting COHORT 2 inclusion criteria, who have BILATERAL "severe lower extremity injuries".
   * COHORT 2C (ACS GROUP): Patients meeting COHORT 2 inclusion criteria, who have been clinically diagnosed by the treating provider using that treating provider's standards of diagnosing ACS and the patient, in addition to being diagnosed with ACS, undergoes four-compartment leg fasciotomy. Patients in this cohort need data collection to start BEFORE fasciotomy and continue AFTER fasciotomy.
2. Record provider comments regarding usability of the technology in its new embodiment and areas of needed design improvement. Apply this knowledge to perfect the industrial design and functionality of the final device.
3. Establish evidenced-based clinical guidelines for the diagnosis and management of ACS in traumatically injured soldiers to be tested in a subsequent interventional clinical (IDE) study.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects
* between the ages of 15 and 65 years old
* (Cohort 1 only) Admitted directly to the ICU of a participating study site
* (Cohort 2 only) Admitted to a participating study site with the following injury/mechanism combinations:

Injuries:

1. Segemental tibia shaft fracture
2. Comminuted tibia shaft fracture
3. Schatzker Type III-VI tibial plateau fractures

Mechanisms:

1. Fall from a height of >= 8 feet
2. Motor vehicle or motorcycle crash
3. Pedestrian versus automobile

Exclusion Criteria:

* Patients, in whom application of NIRS monitoring is viewed as an impediment to care.
* Patients with known prior leg fractures (not related to current injury)
* History of peripheral vascular disease or lower extremity vascular surgery.
* Amputation
* Diagnoses with ACS prior to enrollment
* Spinal injuries resulting in complete loss of function
* Mangled lower extremity
* Bilateral upper extremity injuries

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically injured patients (Cohort 1) or patients with severe lower extremity injuries (Cohort 2), admitted to one of the participating sites, who meet the eligibility criteria described below.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute compartment syndrome (ACS) | 24-48 hours at study site
  The "gold standard" criterion for ACS will be "clinical diagnosis". That is, all subjects undergoing fasciotomy for clinically diagnosed ACS (NOT PROPHYLACTIC fasciotomies) will be considered to have ACS. NIRS values will be compared to clinical diagnosis to determine accuracy and threshold values.

SECONDARY OUTCOMES:
Intracompartmental pressure (ICP) | 24-48 hours at study site
  ICP measurements will be taken at the doctor's discretion, as this is the only existing objective diagnostic tool for ACS. When available, ICP will be compared to NIRS values to assess the magnitude of agreement between the 2 tools.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Freedman, MD, Principal Investigator — Landstuhl Regional Medical Center; William Reisman, MD, Principal Investigator — Emory University; Bruce Ziran, MD, Principal Investigator — Atlanta Medical Center
Locations (2):
- United States (2):
  - Atlanta Medical Center, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia